CLINICAL TRIAL: NCT06386497
Title: Overnight Treatment of Parkinson's Disease Using Vestibular Stimulation From a Rocking Bed (Somnomat Casa) - A Feasibility Study
Brief Title: Acceptability of the Somnomat Casa for the Treatment of Parkinson's Disease
Acronym: Somnomat Casa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-D0100
Record Dates: First submitted 2024-04-15; First posted 2024-04-26 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Vestibular Stimulation; Sleep quality; Rocking bed; Feasibility
MeSH Terms: conditions — Parkinson Disease; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson's disease patients (Experimental): All included Parkinson's disease patients
  Interventions: Device: Nocturnal translational vestibular stimulation

INTERVENTIONS:
Device: Nocturnal translational vestibular stimulation — Nocturnal (overnight) translational vestibular stimulation applied by the rocking bed (Somnomat Casa) for two months in patients familiar home environment.

SUMMARY:
This pilot study aims to evaluate the feasibility and acceptability of nocturnal translational vestibular stimulations (VS) applied by a rocking bed (Somnomat Casa) for two months in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
Twelve PD patients will receive overnight VS in their familiar home environment for two months via the rocking bed. Participants will be given questionnaires to obtain feedback on the acceptability of the nocturnal intervention device.

Effects on sleep, motor and non-motor symptoms, and quality of life will be assessed using the appropriate validated scales and questionnaires. The corresponding assessments will be performed before, during, and two month after the intervention.

Unobtrusive pressure-sensitive textiles and bioradar will be used to record physiological variables such as body position, movements, breathing rate, and heart rate to correlate them to the clinical assessments as well as to markers obtained from actigraphy devices that the patients will be wearing throughout the study.

The primary feasibility outcomes include rate of accrual and retention, adherence to the protocol, acceptability and satisfaction with intervention using rocking bed specific questionnaires, semi-structured interviews, and data collected automatically from the bed.

To assess the preliminary effectiveness of the intervention the secondary outcomes are the change in subjective sleep quality, daytime sleepiness, PD related sleep disorders, mentation, behaviour, mood, activities of daily living, motor performance, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* PD according to the MDS clinical diagnostic criteria for Parkinson's disease
* Suffering from reduced sleep quality as defined by pathological cut-off (score of > 5) on the Pittsburgh Sleep Quality Index (PSQI)
* Patients with stable antiparkinsonian, antidepressant, and sleep medications for six weeks before intervention and maintained on stable medication during the intervention period
* Treatment without bilateral deep brain stimulation
* Fluent in German

Exclusion Criteria:

* Brain disease other than Parkinson's disease (e.g. atypical Parkinsonism, Alzheimer's disease, vascular dementia, multiple sclerosis, stroke, traumatic brain injury, epilepsy, etc.).
* Dementia as defined by a MOCA score lower than 24/30
* Weight > 150kg
* Depression with acute suicidal ideation
* Presence of major ongoing psychiatric illness such as acute non-controlled psychosis
* Poor general health (e.g. non-controlled diabetes, uncontrolled arterial hypertension, therapy for malignancy)
* Inability to follow the procedures of the study, e.g. filling out patient questionnaires due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another interventional trial within the 30 days preceding and during the present study
* Participants with PSQI score lower or equal 5

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of acceptability and feasibility | At Visit 1 (1 month after start of intervention)
  The acceptability and feasibility of the translational vestibular stimulation with the Somnomat Casa will be evaluated with a custom-designed questionnaire. The questionnaire consists of 22 questions including questions with five-point likert scale and open questions ("I fully agree" to "I do not agree at all").
Evaluation of acceptability and feasibility | At Visit 2, at the end of the intervention (after 2 months)
  The acceptability and feasibility of the translational vestibular stimulation with the Somnomat Casa will be evaluated with a custom-designed questionnaire. The questionnaire consists of 22 questions including questions with five-point likert scale and open questions ("I fully agree" to "I do not agree at all").

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | At Baseline Visit (before the intervention)
  The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, assessing a broad range of domains associated with sleep quality, including: usual sleep wake patterns, duration of sleep, sleep latency, the frequency and severity of specific sleep-related problems, and the perceived impact of poor sleep on daytime functioning.
Pittsburgh Sleep Quality Index (PSQI) | At Visit 1 (1 month after start of intervention)
  The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, assessing a broad range of domains associated with sleep quality, including: usual sleep wake patterns, duration of sleep, sleep latency, the frequency and severity of specific sleep-related problems, and the perceived impact of poor sleep on daytime functioning.
Pittsburgh Sleep Quality Index (PSQI) | At Visit 2, at the end of the intervention (after 2 months)
  The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, assessing a broad range of domains associated with sleep quality, including: usual sleep wake patterns, duration of sleep, sleep latency, the frequency and severity of specific sleep-related problems, and the perceived impact of poor sleep on daytime functioning.
Pittsburgh Sleep Quality Index (PSQI) | At Final Visit (two months after the intervention)
  The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, assessing a broad range of domains associated with sleep quality, including: usual sleep wake patterns, duration of sleep, sleep latency, the frequency and severity of specific sleep-related problems, and the perceived impact of poor sleep on daytime functioning.
Epworth Sleepiness Scale (ESS) | At Baseline Visit (before the intervention)
  The ESS is a short self-administered questionnaire designed to assess daytime sleepiness. This basic test involves a self-assessment of how likely a person is to fall asleep in eight different situations.
Epworth Sleepiness Scale (ESS) | At Visit 1 (1 month after start of intervention)
  The ESS is a short self-administered questionnaire designed to assess daytime sleepiness. This basic test involves a self-assessment of how likely a person is to fall asleep in eight different situations.
Epworth Sleepiness Scale (ESS) | At Visit 2, at the end of the intervention (after 2 months)
  The ESS is a short self-administered questionnaire designed to assess daytime sleepiness. This basic test involves a self-assessment of how likely a person is to fall asleep in eight different situations.
Epworth Sleepiness Scale (ESS) | At Final Visit (two months after the intervention)
  The ESS is a short self-administered questionnaire designed to assess daytime sleepiness. This basic test involves a self-assessment of how likely a person is to fall asleep in eight different situations.
Parkinson's Disease Sleep Scale version 2 (PDSS-2) | At Baseline Visit (before the intervention)
  The PDSS-2 is a patient-completed clinical rating scale that assesses the frequency of sleep disturbances over the past week. The PDSS-2 covers three domains: motor symptoms at night, PD specific symptoms at night and disturbed sleep.
Parkinson's Disease Sleep Scale version 2 (PDSS-2) | At Visit 1 (1 month after start of intervention)
  The PDSS-2 is a patient-completed clinical rating scale that assesses the frequency of sleep disturbances over the past week. The PDSS-2 covers three domains: motor symptoms at night, PD specific symptoms at night and disturbed sleep.
Parkinson's Disease Sleep Scale version 2 (PDSS-2) | At Visit 2, at the end of the intervention (after 2 months)
  The PDSS-2 is a patient-completed clinical rating scale that assesses the frequency of sleep disturbances over the past week. The PDSS-2 covers three domains: motor symptoms at night, PD specific symptoms at night and disturbed sleep.
Parkinson's Disease Sleep Scale version 2 (PDSS-2) | At Final Visit (two months after the intervention)
  The PDSS-2 is a patient-completed clinical rating scale that assesses the frequency of sleep disturbances over the past week. The PDSS-2 covers three domains: motor symptoms at night, PD specific symptoms at night and disturbed sleep.
Restless Legs Syndrome Rating Scale (IRLS) | At Baseline Visit (before the intervention)
  IRLS is a 10-item questionnaire to assess the severity of the Restless Legs Syndrome (RLS).
Restless Legs Syndrome Rating Scale (IRLS) | At Visit 1 (1 month after start of intervention)
  IRLS is a 10-item questionnaire to assess the severity of the Restless Legs Syndrome (RLS).
Restless Legs Syndrome Rating Scale (IRLS) | At Visit 2, at the end of the intervention (after 2 months)
  IRLS is a 10-item questionnaire to assess the severity of the Restless Legs Syndrome (RLS).
Restless Legs Syndrome Rating Scale (IRLS) | At Final Visit (two months after the intervention)
  IRLS is a 10-item questionnaire to assess the severity of the Restless Legs Syndrome (RLS).
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | At Baseline Visit (before the intervention)
  The MDS-UPDRS is a scale used to measure the severity of PD. A higher score denotes greater disability. It includes four parts: mentation, behaviour and mood (MDS-UPDRS I); activities of daily living (MDS-UPDRS II); motor examination MDS-UPDRS III); complication of treatment (MDS-UPDRS IV).
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | At Visit 1 (1 month after start of intervention)
  The MDS-UPDRS is a scale used to measure the severity of PD. A higher score denotes greater disability. It includes four parts: mentation, behaviour and mood (MDS-UPDRS I); activities of daily living (MDS-UPDRS II); motor examination MDS-UPDRS III); complication of treatment (MDS-UPDRS IV).
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | At Visit 2, at the end of the intervention (after 2 months)
  The MDS-UPDRS is a scale used to measure the severity of PD. A higher score denotes greater disability. It includes four parts: mentation, behaviour and mood (MDS-UPDRS I); activities of daily living (MDS-UPDRS II); motor examination MDS-UPDRS III); complication of treatment (MDS-UPDRS IV).
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | At Final Visit (two months after the intervention)
  The MDS-UPDRS is a scale used to measure the severity of PD. A higher score denotes greater disability. It includes four parts: mentation, behaviour and mood (MDS-UPDRS I); activities of daily living (MDS-UPDRS II); motor examination MDS-UPDRS III); complication of treatment (MDS-UPDRS IV).
Parkinson's disease quality of life questionnaire (PDQ-39) | At Baseline Visit (before the intervention)
  The Parkinson's disease quality of life questionnaire evaluates the disease specific QoL. This questionnaire quantifies disease-specific and disease-referred quality of life in PD patients. In 39 items 8 main dimensions are interrogated (mobility, activities of daily living, emotional well-being, stigma, social support, cognitive impairment, communication and bodily discomfort). Each of these 8 domains contributes equally to a summary index of overall disease specific QoL.
Parkinson's disease quality of life questionnaire (PDQ-39) | At Visit 1 (1 month after start of intervention)
  The Parkinson's disease quality of life questionnaire evaluates the disease specific QoL. This questionnaire quantifies disease-specific and disease-referred quality of life in PD patients. In 39 items 8 main dimensions are interrogated (mobility, activities of daily living, emotional well-being, stigma, social support, cognitive impairment, communication and bodily discomfort). Each of these 8 domains contributes equally to a summary index of overall disease specific QoL.
Parkinson's disease quality of life questionnaire (PDQ-39) | At Visit 2, at the end of the intervention (after 2 months)
  The Parkinson's disease quality of life questionnaire evaluates the disease specific QoL. This questionnaire quantifies disease-specific and disease-referred quality of life in PD patients. In 39 items 8 main dimensions are interrogated (mobility, activities of daily living, emotional well-being, stigma, social support, cognitive impairment, communication and bodily discomfort). Each of these 8 domains contributes equally to a summary index of overall disease specific QoL.
Parkinson's disease quality of life questionnaire (PDQ-39) | At Final Visit (two months after the intervention)
  The Parkinson's disease quality of life questionnaire evaluates the disease specific QoL. This questionnaire quantifies disease-specific and disease-referred quality of life in PD patients. In 39 items 8 main dimensions are interrogated (mobility, activities of daily living, emotional well-being, stigma, social support, cognitive impairment, communication and bodily discomfort). Each of these 8 domains contributes equally to a summary index of overall disease specific QoL.
Patients' Global Impression of Severity Scale (PGIS) | At Baseline Visit (before the intervention)
  The Patient Global Impression of Severity scale is a single, self-administered question asking respondents about the severity of their current general condition.
Patients' Global Impression of Change Scale (PGICS) | At Visit 1 (1 month after start of intervention)
  The Patient Global Impression of Change scale is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time.
Patients' Global Impression of Change Scale (PGICS) | At Visit 2, at the end of the intervention (after 2 months)
  The Patient Global Impression of Change scale is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time.
Patients' Global Impression of Change Scale (PGICS) | At Final Visit (two months after the intervention)
  The Patient Global Impression of Change scale is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time.

CONTACTS AND LOCATIONS:
Overall Officials: Lenard Lachenmayer, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Switzerland (2):
  - Insel Gruppe AG, University Hospital Bern, Bern
  - ETH Zurich, Sensory-Motor Systems Lab, IRIS, Zurich

IPD SHARING:
Plan to Share IPD: No